CLINICAL TRIAL: NCT04159454
Title: Pacemaker Induced Transient Dyssynchrony for Treating Heart Failure (PITA-HF): Feasibility, Safety, and Tolerability
Brief Title: PITA-HF: Feasibility, Safety, and Tolerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00220173
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; Dilated Cardiomyopathy
Keywords: Pacing; Heart failure; Dyssynchrony
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: The investigators will inform all subjects initially that 50% of the subjects will have PITA on for the first 8 weeks, and 50% will have PITA on for the last 4 weeks. However, all patients will follow the same protocol consisting of PITA on for Weeks 0-8, and PITA off for Weeks 8-12. Because this is a feasibility, safety, and tolerability trial, there is no need for a placebo or non-treatment group. Each patient serves as his or own control with a period of PITA on and PITA off. This data will help inform the investigators' next studies which will include control groups.
Masking Description: This is a feasibility, safety, and tolerability pilot trial that is double-blinded. To the extent that is possible, the outcome variable collection and analysis will be fully blinded. Only the device nurse responsible for programming ICDs and investigators responsible for performing physical examinations will know specifics of patient protocol (ie which patients will have PITA and when) and will be unblinded; all other investigators and patients will be blinded. Subjects meeting inclusion criteria and not any exclusion criteria (see below) will have PITA on for Weeks 0-8 and PITA off for Weeks 8-12. This design provides assessment of feasibility, tolerability and safety of PITA over a 2 month timepoint and the decay effect of PITA for an additional month once turned off.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PITA Participants (Experimental): All patients in the study are part of the "PITA" arm, where PITA will be on for Weeks 0-8, and off from Weeks 8-12.
  Interventions: Device: PITA

INTERVENTIONS:
Device: PITA — Patients will have PITA turned on to patients' existing Medtronic devices, such that patients will be RV-paced from midnight to 6 AM each night at a rate ~10 beats per minute (BPM) above patients' baseline heart rates during this time period as determined by Holter monitors.

SUMMARY:
Heart failure affects over 25 million people worldwide and nearly 7 million adults in the United States alone. Nearly 25% of patients with heart failure have worsened disease burden from dyssynchronous ventricular contraction due to abnormal electrical impulse propagation. These patients may benefit from cardiac resynchronization therapy (CRT) where contraction between the ventricles is coordinated by simultaneous electrical stimulation of the right and left ventricles. In animal models, CRT changes molecular and cellular biology by improving myofilament function, ion channel regulation, beta-receptor signaling, and overall mitochondrial energetics. In randomized clinical outcomes trials, the use of CRT further reduced the incidence of heart failure events and improved overall mortality. However, nearly 75% of patients with heart failure have synchronous ventricular contraction and therefore do not qualify for CRT. CRT profoundly alters underlying molecular and cellular biology as a result of the transition from dyssynchronous to resynchronized contraction, enhancing myocyte function and adrenergic responsiveness. The investigators previously hypothesized CRT-like benefits could be achieved in otherwise synchronous heart failure by purposely inducing dyssynchrony for several hours each day and then reversing this for the remainder of the time. The investigators termed this pacemaker induced transient dyssynchrony, or PITA, and tested its impact in a canine dilated cardiomyopathy model. Following several weeks of rapid atrial pacing to induce heart failure in the animals, the investigators compared implementing 4-weeks of PITA - consisting of dyssynchronous rapid right ventricular pacing for 6 hours each night and atrial pacing for the remaining time - to animals that always received rapid atrial pacing. The fast rate is used to generate a heart failure phenotype. PITA improved chamber dilation, increased beta-adrenergic responsiveness and contractile function, and improved myofiber structure compared to heart failure canine controls. While first tested in an intact conscious translational model, no study has yet investigated PITA in humans. This pilot research protocol tests the feasibility, safety, and tolerability of PITA in humans with dilated cardiomyopathy. The study will leverage pre-existing Medtronic (Mounds View, MN) pacemaker/defibrillators implanted in dilated cardiomyopathy patients based on current clinical guidelines. If successful, this study will allow for a larger, first-in-human study to assess indexes of left ventricular function in dilated cardiomyopathy patients with PITA.

DETAILED DESCRIPTION:
Over 25 million people worldwide are affected by heart failure. In the United States alone, nearly 7 million adults have heart failure with a prevalence of ~3% of adults over 18 years old. Therapy is directed at the underlying cause of heart failure and stratified by ejection fraction. In patients with heart failure with reduced ejection fraction (HFrEF), standard guideline-directed medical therapy consists, at minimum, of maximally tolerated beta blockade and angiotension converting enzyme (ACE) inhibitor or angiotension receptor blockade (ARB) therapy. Additive therapies may include further neurohormonal blockade with spironolactone or eplerenone, with symptomatic management anchoring on lifestyle modifications and diuretics.

Antiarrhythmic devices are commonly employed in HFrEF patients. Patients with ischemic heart disease and an ejection fraction below 35% are recommended for internal cardiac defibrillators (ICD) as primary prevention, and those who have experienced episodes of sudden cardiac arrest or syncope related to ventricular arrhythmia are candidates for ICDs as secondary prevention. Individuals with non-ischemic HFrEF are recommended for secondary prevention ICD implantation.

Another device therapy is cardiac resynchronization therapy (CRT) used in HFrEF patients with underlying delayed electromechanical conduction delay. With differences in regional electrical propagation as with left bundle branch blocks or intraventricular conduction delays, the left ventricular free wall and septum (left and right sides) contract in a discoordinate manner, reducing overall pump efficiency and mechanoenergetic performance. CRT employs pacing of the left ventricular lateral wall and right ventricular septum simultaneously, recoordinating electromechanical activation to improve ventricular function.

The investigators previously showed that while CRT improves chamber-level mechanoenergetics, it also results in profound molecular and myocyte changes that are often global in nature and underlie functional improvement. In a dilated cardiomyopathy canine model (rapid pacing for 6 weeks), CRT improves myofilament function, ion channel regulation, beta-receptor signaling, and mitochondrial function and energetics. Several of these features have been examined in human endocardial biopsies following CRT supporting the appearance of these features in patients.

Furthermore, in large-scale, randomized trials, CRT improved cardiovascular outcomes. The MIRACLE trial randomized 453 patients to CRT with EF <35% and QRS >130 ms to CRT vs control and found significant improvements in clinical endpoints of six minute walk distance, functional class, quality of life, and ejection fraction. The COMPANION trial randomized 1,520 patients with advanced heart failure and intraventricular conduction delays to standard medical therapy, CRT-P (pacemaker only), or CRT-D (defibrillator). In both CRT groups, there were significant reductions in the primary endpoint of time to death or hospitalization, with relative reductions of 34% and 40% respectively. The MADIT-CRT trial randomized 1,820 patients with ejection fraction <30% and QRS duration of >130 milliseconds with New York Heart Association class I or II symptoms to CRT-D or ICD therapy alone. In the CRT-D group, a significant reduction in the primary endpoint of death from any cause or nonfatal heart failure event was observed. Interestingly, the Echo CRT trial randomized 809 patients with ejection fraction <35%, QRS <130 milliseconds, and New York Heart Association class III or IV heart failure with echocardiographic evidence of left ventricular dyssynchrony to CRT vs dual chamber pacemaker. Unlike MADIT-CRT, there was no significant differences in the primary endpoint of death or first hospitalization for worsening heart failure between the groups prompting the trial to terminate early, suggesting that the benefit from CRT is contingent upon high baseline level of ventricular dyssynchrony. Based on MADIT-CRT and other large-scale trials, CRT is now recommended as per the recent American College of Cardiology/American Heart Association heart failure guidelines as Class I indication in patients with (1) New York Heart Association (NYHA) Class III or IV symptoms despite optimal heart failure therapy with left ventricular ejection fraction (LVEF) <35% and prolonged QRS duration or (2) NYHA Class I, II, or III symptoms with LVEF <50% on optimal heart failure therapy with expected high percentage of ventricular pacing.

Despite the success of CRT as additive therapy, it is limited to a subset of heart failure patients with a wide QRS complex and evidence of mechanical dyssynchrony. The majority of patients (~75%) with HFrEF have synchronous ventricular contraction with narrow QRS complexes on surface ECGs and so do not qualify for CRT. However, the molecular/cellular biology following CRT raised a provocative question: might purposely inducing dyssynchrony in heart failure for a discrete period of time and then reversing it also confer similar benefits to CRT? This notion of purposely applying a stimulus that if done for a prolonged period has adverse impact but more short term and then reversed yields therapeutic benefit has an analogy to ischemic pre-conditioning, where brief exposure to ischemia and then reperfusion instills protective molecular changes to better handle subsequent prolonged ischemic injury.

To test this hypothesis, the investigators first tested the effects of pacemaker-induced transient dyssynchrony (termed PITA) in a dilated cardiomyopathy canine model. After 2-weeks of synchronous atrial tachypacing at 200 beats per minute to induce dilated cardiomyopathy, dogs were exposed to PITA consisting of dyssynchronous (with respect to atrial contraction) right ventricular pacing at the same rate from midnight to 6 AM each day, corresponding to the period of least activity. Pacing was switched to rapid atrial pacing (same rate) for the rest of the day: 6 AM to midnight. A control group of dogs received rapid atrial pacing only. Indices of global left ventricular function and cellular/molecular changes were compared between the groups and to controls without heart failure. The investigators found that intact left ventricular chamber end diastolic and end systolic diameters were smaller and ejection fraction greater in dogs receiving PITA. Left ventricular end diastolic pressure was decreased in the PITA group versus HF controls. Left ventricular contractility also improved in the PITA group, primarily with co-administered dobutamine to stimulate contractile reserve. The latter ultimately achieved levels similar to those in healthy controls, so the adrenergic response improvement was substantial. Thus, PITA attenuated adverse remodeling due to synchronous HF in the intact heart.

At the myocyte level, PITA improved sarcomere shortening, peak calcium transient, myofilament sarcomere function (peak myocyte force-calcium dependence), and beta adrenergic stimulated response (both b1 and b2). Ultrastructurally, PITA preserved myofilament assembly and integrity, and prevented the formation of low-force generating myofibrils. Interestingly, all of these beneficial effects of PITA were only seen when a contiguous period of right ventricular (RV) pacing was applied. When RV pacing was randomly distributed over a 24-hour period, no significant mechanoenergetic or cellular/molecular differences were seen between the treated and control HF groups.

To date, no study has investigated whether similar benefits of PITA are observed in humans with HFrEF. PITA can be easily implemented in HFrEF patients with primary or secondary prevention ICDs or pacemakers inserted to counter bradycardia. Not all pacemaker devices can currently do this, but multiple Medtronic (Mounds View, MN) devices have what is called a Sleep Function feature whereby the pacing rate can be automatically modified during predefined sleep periods, generally lowering this rate so a slower intrinsic non-paced rate occurs. While incorporated to help some patients who felt hearts beat when the patients slept, the feature is in fact rarely used. However, the software has the capacity to be inverted - where the "sleep period" is set to extend from 6 AM to midnight, and then the daytime (faster backup pacing rate) occurs from midnight to 6 AM. The investigators can then pace the RV at a rate that is ~10 bpm above the upper sinus rate observed during the normal sleep hours in a given patient, assuring that there will be dyssynchronous contraction during those hours. In the morning, the rate would fall to below sinus rate to enable normal contraction (synchronous) to be restored.

Given the increasing incidence and prevalence of HFrEF with associated morbidity and mortality, it is important to find additional avenues to intervene and provide beneficial therapies in addition to established medical therapy. While synchronous contraction is a sought-after goal for patients with HFrEF, PITA may be even better and provide an additional device-based therapy to improve heart failure symptoms and overall trajectory in those who already have cardiac defibrillators or meet indications for implantation. Thus, further investigation of the efficacy and safety of these treatments in the HFrEF population without known dyssynchrony is warranted.

This index pilot trial will test the feasibility, safety, and tolerability of PITA in dilated cardiomyopathy patients with low pacing burden to ensure ventricular capture during RV pacing and to enroll patients who otherwise do not meet criteria for CRT. If successful, this will allow subsequent study on changes in left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years of age
* Ejection fraction of <40% by noninvasive testing (TTE, nuclear stress, cardiac MRI) within 6 months of study enrollment
* Presence of Medtronic device (single chamber ICD or dual chamber ICD) with Sleep Function feature (Models: Evera, Maximo II, Virtuoso II, Secura, Protecta)
* Low pacing burden, defined as <5% RV pacing in the prior month as determined by baseline device interrogation (prior to Week 0)
* Narrow QRS complex (<100 milliseconds) on baseline ECG without any pacing or with atrial pacing only
* No evidence of incomplete bundle branch block or intraventricular conduction delay, defined as QRS 100-120 milliseconds with: a. S wave in V1 with broad R waves in I, aVL, and V6 b. RSR' in v1 with terminal S waves in I, aVL, and V6 c. not meeting patterns in a or b but with QRS complex 100-120 milliseconds
* No indications for CRT-D upgrade at time of enrollment
* Followed by a physician for treatment of heart failure
* Currently receiving guideline-directed medical therapy for HFrEF
* No changes in diuretic over the past 30 days
* Willingness to provide informed consent
* Negative pregnancy test in a female of child bearing potential

Exclusion Criteria:

* Age <18 years
* Ejection fraction >40% by noninvasive testing in the preceding 12 months
* Acute coronary syndrome within 4 weeks as defined by electrocardiographic (ECG) ST-segment depression or prominent T-wave inversion and/or positive biomarkers of necrosis (e.g., troponin) in the absence of ST-segment elevation and in an appropriate clinical setting (chest discomfort or anginal equivalent)
* Hospital admission for acute decompensated heart failure in the prior 30 days
* Non-Medtronic implanted device or Medtronic device lacking Sleep Function, or Medtronic pacemaker without ICD
* High pacing burden defined as >5% right ventricular pacing in the preceding month based on interrogation
* Meets indication for CRT-D upgrade at the time of enrollment
* Not currently on guideline-directed therapy or non-compliant with medical therapy, assessed through patient interview and review of medical charts
* Non-compliant with medical visits defined as >3 missed clinical visits in the prior year
* NYHA Class IV symptoms at time of enrollment
* Hemodynamically significant arrhythmias including supraventricular tachycardias not responsive to rate control therapies or resulting in hemodynamic instability, sustained ventricular tachycardia (defined as >30 seconds of VT), or defibrillator shock within 4 weeks
* Cardiac arrest within the prior 6 months
* Coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) within the prior 3 months, or recent coronary angiogram with plans for CABG or PCI (unrevascularized disease)
* Presence of durable mechanical hemodynamic support (left ventricular assist device)
* Actively listed for cardiac transplantation, prior history of cardiac transplantation or undergoing evaluation for cardiac transplantation
* Actively listed for any other organ transplantation or undergoing evaluation for any other organ transplantation
* Planned surgical intervention in the next 1 year
* History of persistent, permanent, or long-standing atrial fibrillation
* Terminal illness (other than HF) with expected survival of less than 1 year
* Other end-organ, permanent dysfunction including severe chronic obstructive pulmonary disease (COPD) by Gold's criteria or severe pulmonary disease requiring oxygen, cirrhosis of any cause, renal failure on dialysis, chronic untreatable infectious disease, underlying malignancy undergoing active treatment (chemotherapy, radiation therapy, planned surgical resection of tumor), uncontrolled endocrinologic disorder (thyroid dysfunction, adrenal disease, etc.) requiring ongoing medication titration
* Previous symptomatic intolerance to right ventricular pacing
* Enrollment or planned enrollment in another randomized clinical trial
* Inability to comply with planned study procedures
* Pregnancy or nursing mothers, or women planning on becoming pregnant
* Irreversible neurologic function with inability to provide own consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by percent ventricular capture through Holter monitoring | Up to 7 weeks
  Patients will be given 48-hour Holter monitors at Week 1, Week 4, and Week 7. The average heart rate in beats per minute (bpm) during sleep hours (midnight-6 AM) will be recorded. Percent ventricular capture will be defined as the percentage of heart rate during this time period that is above the pre-specified heart rate set for each patient during the "sleep" period. Percent will be defined from 0-100%, with the latter indicating all ventricular beats are paced from the right ventricle, and the former indicating that no ventricular beats are paced.
Safety as assessed by number of arrhythmia episodes via device interrogation | Up to 3 months
  Patients will have patient's ICD devices interrogated throughout the study as per the study protocol, and the number of sustained ventricular tachycardia (VT) episodes, non-sustained VT episodes, and ventricular fibrillation (VF) episodes will be counted and recorded. At the conclusion of each interrogation, the device counter will be reset such that the next interrogation is only reflective of the interim time period.
Safety as assessed by the number of hospitalizations or ER visits for arrhythmia or heart failure | Up to 3 months
  As per the study protocol, patient interviews and chart reviews will be implemented to count the number of ER visits or hospitalizations for issues related to arrhythmia or clinical heart failure decompensation.
Tolerability as assessed by change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Baseline, Week 4, Week 8 and Week 12
  Patients will fill out the Kansas City Cardiomyopathy Questionnaire at Weeks 0, 4, 8, and 12, and a numerical score is provided at each timepoint and compared. Scores are from 0-100, with higher scores corresponding to improved quality of life and associated with New York Heart Association Class I symptoms, and lower scores associated with poorer quality of life and association with New York Heart Association Class IV symptoms.
Tolerability as assessed by change in distance during 6-minute walk test | Baseline and Week 8
  Distance (feet) during 6 minute-walk test will be obtained and recorded at Weeks 0 and 8. Larger distances are associated with improved functional status/capacity. Typical distances covered in healthy individuals range from 1300-2300 ft.
Safety as assessed by number of tachytherapies delivered by ICDs | Up to 3 months
  Patients will have patient's ICD devices interrogated throughout the study as per the study protocol, and the number of tachytherapies delivered (ATP or ICD shocks) will be counted and recorded. At the conclusion of each interrogation, the device counter will be reset such that the next interrogation is only reflective of the interim time period.
Tolerability as assessed by change in Global Well-Being score on a Visual Analog Scale | Baseline, Week 4, Week 8 and Week 12
  Patients will fill out the Global Well-Being score at Weeks 0, 4, 8, and 12, and a numerical score is provided at each timepoint and compared. The scale is from 0-100, with higher numbers corresponding to improved well-being, and lower numbers corresponding to lower well-being.
Tolerability as assessed by change in Subjective Dyspnea score on a Visual Analog Scale | Baseline, Week 4, Week 8 and Week 12
  Patients will fill out the Subjective Dyspnea score at Weeks 0, 4, 8, and 12, and a numerical score is provided at each timepoint and compared. The score is from 0-100, with higher scores indicating improved subjective dyspnea, and lower scores indicating worsened subjective dyspnea.
Tolerability as assessed by change in Frailty Index | Baseline, Week 4, Week 8 and Week 12
  The Frailty Index will be assessed by the Johns Hopkins Older Americans Independence Center Online Frailty Assessment Tool. Patients will by assessed by the Frailty Index at Weeks 0, 4, 8, and 12, and a numerical score is provided at each timepoint and compared. The score is from 0-5, indicating frail (score 3-5), pre-frail (score 1 or 2) or robust (score 0).
Tolerability as assessed by change in Sleep Quality | Baseline, Week 1, Week 4, Week 5, Week 8 and Week 12
  Sleep Quality will be assessed by Pittsburgh Sleep Quality Index (PSQI). Patients will fill out the Pittsburgh Sleep Quality Index at Weeks 0, 1, 4, 5, 8, and 12, and a numerical score is provided at each timepoint and compared. Scores range from 0-21, with lower scores corresponding to healthier sleep habits and improved sleep quality, and higher scores corresponding to worsened sleep quality.

SECONDARY OUTCOMES:
Presence of dyssynchrony on echocardiography | Baseline, Week 8
  Dyssynchrony will be determined by differences in right and left ventricle contraction and regional wall contraction differences in the left ventricle using echocardiography. It will be reported as present or not per participant.
  Echocardiograms will be obtained at Weeks 0 and 8. To assess interventricular dyssynchrony, onset of QRS complex to peak pulmonic valve inflow or peak aortic valve inflow >40 ms or aortic pre-ejection delay >140 ms is considered significant. To assess intraventricular or LV mechanical dyssynchrony, M-mode in the parasternal long axis will be used to assess septal to posterior wall motion delay, with values >130 ms considered significant. Furthermore, time to onset or time to peak systolic velocity of 4 opposing walls >65 ms is considered significant, and will be obtained from parasternal short axis views of the LV via tissue doppler.
Change in N-terminal pro b-type natriuretic peptide (NT pro-BNP) values | Baseline, Week 4 and Week 12
  NT pro-BNP values (pg/mL) will be obtained at Weeks 0, 4, and 12 and be compared. Values less than 125 pg/mL are considered normal.
Change in troponin values (ng/mL) | Baseline, Week 4 and Week 12
  Troponin values (ng/mL) will be obtained at Weeks 0, 4, and 12 and be compared. Values less than 0.04 ng/mL are considered normal.
Change in sodium values (mEq/L) | Baseline, Week 4 and Week 12
  Changes in sodium volume (mEq/L) will be obtained at Weeks 0, 4, and 12 and be compared. Values 135-145 mEq/L are considered normal.
Change in serum creatinine values (mg/dL) | Baseline, Week 4 and Week 12
  Serum creatinine values (mg/dL) will be obtained at Weeks 0, 4, and 12 and be compared. Values less than 1.2 mg/dL are considered normal.
Change in serum blood urea nitrogen (BUN) values | Baseline, Week 4 and Week 12
  Serum BUN values (mg/dL) will be obtained at Weeks 0, 4, and 12 and be compared. Values 7 to 20 mg/dL are considered normal.

OTHER OUTCOMES:
Change in left ventricular (LV) chamber dimensions | Baseline, Week 8
  Change in LV chamber dimensions (systolic and diastolic dimension in centimeters) as measured via the parasternal long-axis view as part of standard echocardiography at Week 0 and Week 8. Diastolic dimensions less than 6 cm and systolic dimensions less than 4 cm are considered normal.
Change in left ventricular (LV) ejection fraction | Baseline, Week 8
  Changes in LV ejection fraction (as a percentage) measured via method of discs via the 4-chamber apical echocardiogram view and the 2-chamber echocardiogram view at Week 0 and Week 8. Ejection fractions of 52-65% are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Sharma, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirk JA, Chakir K, Lee KH, Karst E, Holewinski RJ, Pironti G, Tunin RS, Pozios I, Abraham TP, de Tombe P, Rockman HA, Van Eyk JE, Craig R, Farazi TG, Kass DA. Pacemaker-induced transient asynchrony suppresses heart failure progression. Sci Transl Med. 2015 Dec 23;7(319):319ra207. doi: 10.1126/scitranslmed.aad2899. PMID 26702095
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Background] Shen L, Jhund PS, McMurray JJV. Declining Risk of Sudden Death in Heart Failure. N Engl J Med. 2017 Nov 2;377(18):1794-5. doi: 10.1056/NEJMc1711901. No abstract available. PMID 29091558
- [Background] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701
- [Background] Kirk JA, Kass DA. Cellular and Molecular Aspects of Dyssynchrony and Resynchronization. Heart Fail Clin. 2017 Jan;13(1):29-41. doi: 10.1016/j.hfc.2016.07.003. PMID 27886930
- [Background] Chakir K, Depry C, Dimaano VL, Zhu WZ, Vanderheyden M, Bartunek J, Abraham TP, Tomaselli GF, Liu SB, Xiang YK, Zhang M, Takimoto E, Dulin N, Xiao RP, Zhang J, Kass DA. Galphas-biased beta2-adrenergic receptor signaling from restoring synchronous contraction in the failing heart. Sci Transl Med. 2011 Sep 14;3(100):100ra88. doi: 10.1126/scitranslmed.3001909. PMID 21918105
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Ruschitzka F, Abraham WT, Singh JP, Bax JJ, Borer JS, Brugada J, Dickstein K, Ford I, Gorcsan J 3rd, Gras D, Krum H, Sogaard P, Holzmeister J; EchoCRT Study Group. Cardiac-resynchronization therapy in heart failure with a narrow QRS complex. N Engl J Med. 2013 Oct 10;369(15):1395-405. doi: 10.1056/NEJMoa1306687. Epub 2013 Sep 2. PMID 23998714
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Heart Rhythm Society. 2012 ACCF/AHA/HRS focused update incorporated into the ACCF/AHA/HRS 2008 guidelines for device-based therapy of cardiac rhythm abnormalities: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. Circulation. 2013 Jan 22;127(3):e283-352. doi: 10.1161/CIR.0b013e318276ce9b. Epub 2012 Dec 19. No abstract available. PMID 23255456
- [Background] Curtis AB, Worley SJ, Adamson PB, Chung ES, Niazi I, Sherfesee L, Shinn T, Sutton MS; Biventricular versus Right Ventricular Pacing in Heart Failure Patients with Atrioventricular Block (BLOCK HF) Trial Investigators. Biventricular pacing for atrioventricular block and systolic dysfunction. N Engl J Med. 2013 Apr 25;368(17):1585-93. doi: 10.1056/NEJMoa1210356. PMID 23614585
- [Background] Aiba T, Hesketh GG, Barth AS, Liu T, Daya S, Chakir K, Dimaano VL, Abraham TP, O'Rourke B, Akar FG, Kass DA, Tomaselli GF. Electrophysiological consequences of dyssynchronous heart failure and its restoration by resynchronization therapy. Circulation. 2009 Mar 10;119(9):1220-30. doi: 10.1161/CIRCULATIONAHA.108.794834. Epub 2009 Feb 23. PMID 19237662
- [Background] Chen CH, Fetics B, Nevo E, Rochitte CE, Chiou KR, Ding PA, Kawaguchi M, Kass DA. Noninvasive single-beat determination of left ventricular end-systolic elastance in humans. J Am Coll Cardiol. 2001 Dec;38(7):2028-34. doi: 10.1016/s0735-1097(01)01651-5. PMID 11738311
- [Background] Khurshid S, Epstein AE, Verdino RJ, Lin D, Goldberg LR, Marchlinski FE, Frankel DS. Incidence and predictors of right ventricular pacing-induced cardiomyopathy. Heart Rhythm. 2014 Sep;11(9):1619-25. doi: 10.1016/j.hrthm.2014.05.040. Epub 2014 Jun 2. PMID 24893122
- [Background] Link MS, Hellkamp AS, Estes NA 3rd, Orav EJ, Ellenbogen KA, Ibrahim B, Greenspon A, Rizo-Patron C, Goldman L, Lee KL, Lamas GA; MOST Study Investigators. High incidence of pacemaker syndrome in patients with sinus node dysfunction treated with ventricular-based pacing in the Mode Selection Trial (MOST). J Am Coll Cardiol. 2004 Jun 2;43(11):2066-71. doi: 10.1016/j.jacc.2003.10.072. PMID 15172414
- [Background] Morris-Thurgood JA, Frenneaux MP. Pacing in congestive heart failure. Curr Control Trials Cardiovasc Med. 2000;1(2):107-114. doi: 10.1186/cvm-1-2-107. PMID 11714422